CLINICAL TRIAL: NCT00499967
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled Assessment of the Safety, Tolerability, and Activity of GS-9191 Ointment for the Treatment of External Genital and Perianal Warts Caused by Human Papilloma Virus Infection
Brief Title: Safety and Effectiveness Study of an Experimental Topical Ointment (GS-9191) for the Treatment of Genital Warts
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Elsa Mondou, MD, Gilead Sciences, Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GS-US-197-0101
Record Dates: First submitted 2007-07-10; First posted 2007-07-12 (Estimated); Last update posted 2009-04-09 (Estimated); Status verified 2009-04

CONDITIONS: Genital Warts
Keywords: genital warts; venereal warts; human papilloma virus
MeSH Terms: conditions — Condylomata Acuminata | interventions — GS-9191

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Cohort 1 (Experimental): GS-9191 0.01% ointment
  Interventions: Drug: GS-9191 ointment
- Cohort 2 (Experimental): GS-9191 0.03% ointment
  Interventions: Drug: GS-9191 ointment
- Cohort 3 (Experimental): GS-9191 0.1% ointment
  Interventions: Drug: GS-9191 ointment
- Cohort 4 (Active Comparator): GS-9191 0.3%
  Interventions: Drug: GS-9191
- Cohort 5 (Active Comparator): GS-9191 1.0%
  Interventions: Drug: GS-9191
- Cohorts 1, 2, 3, 4 & 5 (Placebo Comparator): Placebo in all cohorts
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GS-9191 ointment — GS-9191 ointment (0.01%, 0.03%, or 0.1%) or placebo applied topically to anogenital warts for one or three cycles, each cycle lasting 5 consecutive nights of ointment application followed by 9 nights off-ointment. The strength of GS-9191 ointment is cohort-dependent, with escalation to higher dose cohorts dependent upon safety and tolerability in the previous cohort.
  Arms: Cohort 1; Cohort 2; Cohort 3
Drug: GS-9191 — GS-9191 ointment (0.3% or 1.0%) or placebo applied topically to anogenital warts for one or three cycles; each cycle consists of dosing occuring over a 5-night period with ointment application on nights 1, 3 and 5 followed by a 9-day off-ointment period. The strength of GS-9191 ointment is cohort-dependent, with escalation to higher dose cohorts dependent upon safety and tolerability in the previous cohort.
  Arms: Cohort 4; Cohort 5
Drug: Placebo — Placebo matching GS-9191 ointment
  Arms: Cohorts 1, 2, 3, 4 & 5

SUMMARY:
The purpose of this study is to assess the safety, tolerability and activity of GS-9191 ointment in the treatment of genital warts. GS-9191 ointment is intended for topical application directly to genital warts on the skin.

ELIGIBILITY:
Inclusion Criteria:

* Have 2 or more genital warts of prespecified sizes on external surfaces of the body.
* If HIV positive, have HIV RNA < 400 copies/mL, CD4 count of ≥ 400 cells/mm3, and be taking a triple combination antiviral medication regimen

Exclusion Criteria:

* Prior genital wart treatment within 8 weeks
* Pregnancy or breast-feeding
* Presence of broken or non-intact skin near the wart site or other skin disease at the wart site (e.g., herpes genitalis)
* Treatment with systemic steroids, systemic immunomodulators, immunosuppressants, or chemotherapeutic agents within 3 months
* Current or prior diagnosis of Bowenoid papulosis, cancer, or pre-cancerous tissue in the genital area

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 202 (Actual)
Dates: Start 2007-08; Primary Completion 2009-02 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Regression of anogenital warts based on the total surface area involved by treated warts before, during, and after treatment. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Elsa Mondou, MD, Study Director — Gilead Sciences
Locations (23):
- United States (23):
  - Tucson, Arizona
  - Beverly Hills, California
  - Mission Viejo, California
  - San Francisco, California
  - Santa Rosa, California
  - Vallejo, California
  - Orlando, Florida
  - Tampa, Florida
  - Indianapolis, Indiana
  - St Louis, Missouri
  - Las Vegas, Nevada
  - New York, New York
  - Stony Brook, New York
  - Raleigh, North Carolina
  - Tulsa, Oklahoma
  - Portland, Oregon
  - Greenville, South Carolina
  - Chattanooga, Tennessee
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Seattle, Washington